CLINICAL TRIAL: NCT05819112
Title: A Comparison of Extended Versus Conventional Duration of Enoxaparin Prophylaxis for VTE and Bleeding Event Risk in a Population With Acute Medical Illness
Brief Title: A Comparison of Extended Versus Conventional Duration of Enoxaparin Prophylaxis (i.e., Preventive Treatment) for Venous Thromboembolism (VTE, i.e., Blood Clots in the Veins) and Bleeding Event Risk in a Population With Acute Medical Illness
Status: Terminated | Type: Observational
Why Stopped: Sponsor's decision. Termination decision unrelated to safety profile.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: PDE0093; U1111-1288-8339 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional prophylaxis: Participants hospitalized for acute medical illness receiving conventional (i.e., once daily for 7 days) enoxaparin VTE prophylaxis
- Extended prophylaxis: Participants hospitalized for acute medical illness receiving extended duration (i.e., once daily for 14, 21 or 28 days) enoxaparin VTE prophylaxis

SUMMARY:
Venous Thromboembolism (VTE), including deep vein thrombosis (DVT) and pulmonary embolism (PE), is associated with an increase in risk of mortality and long-term disability and is a major contributor to global disease burden. Participants hospitalized with an acute medical illness are at increased risk of VTE.

This study a non-interventional study which analyzes data already collected in the Optum US clinical database. Its aim is to compare conventional versus extended duration prophylaxis with enoxaparin on the incidence of VTE and bleeding events in participants hospitalized for acute medical illness. The first date of enoxaparin treatment will be the index date.

DETAILED DESCRIPTION:
The study population will be developed from the Optum Clinical database in the United States, representing routine clinical practice. Study population will comprise of participants hospitalized for an acute medical illness receiving enoxaparin during hospitalization. The first date of enoxaparin treatment will be the index date. The study period will be from February 2010 to September 2021. Participants will be followed for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for the following acute conditions:

  * Infection
  * Respiratory insufficiency
  * Inflammatory condition
  * Cancer
  * Heart failure
  * Ischemic stroke
* Initiation of enoxaparin prophylaxis during hospitalization (index date)
* Age ≥40 years

Exclusion Criteria:

* Symptomatic VTE or major bleeding event 90-days prior to index date
* Major surgery within (+1,-90) days from index date
* Ongoing anticoagulation therapy (medication supply within [-2,-32] days from index date)
* Atrial fibrillation
* Chronic kidney disease (CKD) stages IV and V, or dialysis

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants hospitalized for an acute medical illness receiving enoxaparin during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 14799 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in the incidence of VTE, from index date to Day 90 | Retrospective data analysis from February, 2010 to September, 2021, with this endpoint evaluated up to 90 days after the individual participant's index date.
  VTE event will be identified via an algorithm based on the International Classification of Disease-10th revision and 9th revision (ICD-10 and ICD-9) codes.
Change in the incidence of major bleeding, from index date to Day 90 | Retrospective data analysis from February, 2010 to September, 2021, with this endpoint evaluated up to 90 days after the individual participant's index date.
  Major bleeding event will be identified via an algorithm based on the International Classification of Disease-10th revision and 9th revision (ICD-10 and ICD-9) codes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi U.S., Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org